CLINICAL TRIAL: NCT03549442
Title: Phase 1 Study of CART-BCMA With or Without huCART19 as Consolidation of Standard First or Second-Line Therapy for High-Risk Multiple Myeloma
Brief Title: Up-front CART-BCMA With or Without huCART19 in High-risk Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 828773
Record Dates: First submitted 2018-04-27; First posted 2018-06-08 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; BCMA CART; huCART19
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Three separate phases. Phases A and C are non-randomized, Phase B is randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase A (Experimental): Safety Run-in to test the safety of CART-BCMA + huCART19 as split-dose infusions after lymphodepleting chemotherapy with cyclophosphamide + fludarabine in patients who have relapsed/refractory myeloma after two prior regimens but who are responding to their current therapy.
  Interventions: Combination Product: BCMA CART + huCART19
- Phase B (Experimental): Randomization Phase in which patients responding to first or second-line therapy will receive either CART-BCMA alone (Cohort 1) or CART-BCMA + huCART19 (Cohort 2) as split-doses after lymphodepleting chemotherapy with cyclophosphamide + fludarabine.
  Interventions: Combination Product: CART BCMA or CART BCMA + huCART19
- Phase C (Experimental): Single-dose infusion phase to test the safety of single-dose infusion of CART-BCMA alone (Cohort 1) and CART-BCMA + huCART19 (Cohort 2) as single-dose infusions after lymphodepleting chemotherapy with cyclophosphamide + fludarabine in patients responding to first- or second-line therapy.
  Interventions: Combination Product: Single-dose infusion of CART BCMA or CART BCMA + huCART19
- Phase A Expansion (Experimental): Once safety of CART-BCMA/huCART19 combination therapy is established in Phase A, an expansion of Phase A will occur in which the Phase A target population (patients with relapsed/refractory multiple myeloma responding to a standard salvage therapy regimen) will receive both CART-BCMA and huCART19. Enrollment into the Phase A Expansion may occur concurrently with Phase B once opened.
  Interventions: Combination Product: BCMA CART + huCART19

INTERVENTIONS:
Combination Product: BCMA CART + huCART19 — The target dose for CART-BCMA and huCART19 will be 5x108 CAR-expressing cell for each product. Split dose infusions will consist of a 10% dose (of one or both products) on the first infusion day, 30% dose (of one or both products) on the second infusion day, or 60% dose (of one or both products) on the third infusion day. Infusion days may be spread over 7 calendar days due to scheduling constraints or to allow observation of suspected early cytokine release syndrome or other toxicity. Infusions will begin 3 days (+/- 1 day) after completion of lymphodepleting chemotherapy with cyclophosphamide + fludarabine.
  Arms: Phase A
Combination Product: CART BCMA or CART BCMA + huCART19 — The target dose for CART-BCMA and huCART19 will be 5x108 CAR-expressing cell for each product. Cohort 1 refers to the group of subjects assigned to receive CART-BCMA alone; Cohort 2 refers to the group of subjects assigned to receive CART-BCMA + huCART19. Split dose infusions will consist of a 10% dose (of one or both products) on the first infusion day, 30% dose (of one or both products) on the second infusion day, or 60% dose (of one or both products) on the third infusion day. Infusion days may be spread over 7 calendar days due to scheduling constraints or to allow observation of suspected early cytokine release syndrome or other toxicity. Infusions will begin 3 days (+/- 1 day) after completion of lymphodepleting chemotherapy with cyclophosphamide + fludarabine.
  Arms: Phase B
Combination Product: Single-dose infusion of CART BCMA or CART BCMA + huCART19 — The target dose for CART-BCMA and huCART19 will be 5x108 CAR-expressing cell for each product. Cohort 1 refers to the group of subjects assigned to receive single dose infusions of CART-BCMA alone; Cohort 2 refers to the group of subjects assigned to receive single dose infusions of CART-BCMA + huCART19. Infusions will begin 3 days (+/- 1 day) after completion of lymphodepleting chemotherapy with cyclophosphamide + fludarabine.
  Arms: Phase C
Combination Product: BCMA CART + huCART19 — The target dose for CART-BCMA and huCART19 will be 5x108 CAR-expressing cell for each product. Split dose infusions will consist of a 10% dose (of one or both products) on the first infusion day, 30% dose (of one or both products) on the second infusion day, or 60% dose (of one or both products) on the third infusion day. Infusion days may be spread over 7 calendar days due to scheduling constraints or to allow observation of suspected early cytokine release syndrome or other toxicity. Infusions will begin 3 days (+/- 1 day) after completion of lymphodepleting chemotherapy with cyclophosphamide + fludarabine.
  Arms: Phase A Expansion

SUMMARY:
This is an open-label phase 1 study to assess the safety and pharmacodynamics of CART-BCMA, with or without huCART19, in patients responding to first- or second-line therapy for high-risk multiple myeloma. The regimen evaluated in this study is based on established safety of CARTBCMA demonstrated in UPCC 14415/IRB#822756 at dose of 5x108 cells, administered as split infusions, following cyclophosphamide 1.5 g/m2 in patients with relapsed/refractory myeloma. This study tests CART-BCMA (1) as consolidation of early therapy for multiple myeloma, (2) with addition of fludarabine to the lymphodepleting chemotherapy regimen, (3) in combination with huCART19, and (4) as a single rather than split-dose infusion.

DETAILED DESCRIPTION:
Phase A: Safety Run-in to test the safety of CART-BCMA + huCART19 as split-dose infusions after lymphodepleting chemotherapy with cyclophosphamide + fludarabine in patients who have relapsed/refractory myeloma after two prior regimens but who are responding to their current therapy. Phase A Expansion: To occur once safety is demonstrated in Phase A. - Phase B: Randomization Phase in which patients responding to first or second-line therapy will receive either CART-BCMA alone (Cohort

1) or CART-BCMA + huCART19 (Cohort 2) as split-dose infusions after lymphodepleting chemotherapy with cyclophosphamide + fludarabine. Phase C: Single-dose infusion phase to test the safety of single-dose infusion of CART-BCMA alone (Cohort 1) and CART-BCMA + huCART19 (Cohort 2) as single-dose infusions after lymphodepleting chemotherapy with cyclophosphamide + fludarabine in patients responding to first- or second-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a diagnosis of multiple myeloma according to IMWG 2014 criteria106 with any of the following high-risk features. Subjects in the Phase A Expansion are not required to have any high-risk features.

   1. Beta-2-microglobulin ≥ 5.5 mg/L and LDH greater than upper limit of normal. Note: subjects in whom LDH and/or Beta-2-microglobulin were not measured prior to initiation of systemic therapy may qualify based on measurements obtained after initiation of systemic therapy.
   2. High-risk FISH features: at least one of the following [deletion 17p, t(14;16), t(14;20), t(4;14)] in conjunction with Beta-2-microglobulin ≥ 5.5 mg/L (i.e., revised ISS stage 3). Note: subjects in whom Beta-2-microglobulin was not measured prior to initiation of systemic therapy may qualify based on measurements obtained after initiation of systemic therapy.
   3. Metaphase karyotype with >3 structural abnormalities except hyperdiploidy
   4. Plasma cell leukemia (>20% plasma cells in peripheral blood) at any time prior to physician-investigator confirmation of eligibility.
   5. Failure to achieve partial response or better (by IMWG 2016 criteria1) to initial therapy with an "imid/PI" combination (thalidomide, lenalidomide, or pomalidomide in combination with bortezomib, ixazomib, or carfilzomib).
   6. Early progression on first-line therapy, defined as progression (according to IMWG 2016 criteria1)

   i. Within one year of starting first-line therapy with an "imid/PI"combination ii. Within six months of completing first line therapy with an "imid/PI"combination (i.e. a patient who receives an "imid/PI" combination, transitions to observation or maintenance therapy, and progresses within six months of this transition) iii. Within one year of a high-dose melphalan and autologous stem cell transplantation (Phase A subjects only)
2. Subjects must meet the following criteria with respect to prior myeloma therapy:

   a. Phase A and Phase A expansion:

   a. Subjects must meet the following criteria with respect to prior multiple myeloma therapy: i. have disease that has relapsed after or has been refractory to at least two regimens, including a proteasome inhibitor and thalidomide analog (thalidomide, lenalidomide, pomalidomide), OR ii. have disease that has relapsed after or has been refractory to one prior regimen if their prior/current therapy collectively has included all of the following: an "imid/PI" combination, pomalidomide, lenalidomide, daratumumab, and carfilzomib.

   Note: Refractoriness is defined as disease progression on-therapy or within 60 days of stopping therapy.

   b. Subjects must have achieved at least a minimal response (as defined by IMWG 2016 criteria1) to their current regimen.

   c. Subjects must not have received prior treatment with anti-BCMA cellular therapy. Subjects may have received treatment with other BCMA-directed agents (e.g., anti-BCMA antibody-drug conjugates or bispecific antibodies).

   b. Phases B and C:
   1. Subjects must be in their first line of multiple myeloma therapy, with the following exception: subjects who have advanced to second-line therapy due to disease progression during first-line therapy are eligible if such progression occurred within six months of beginning first-line therapy. Lines of therapy are defined by IMWG 2016 criteria1.
   2. Subjects must not have received cytotoxic chemotherapy (e.g., doxorubicin, cyclophosphamide, etoposide, cisplatin) with the following exceptions:

   i. Low-dose weekly cyclophosphamide (≤500 mg/m2/week) ii. Continuous infusion cyclophosphamide, if limited to a single cycle. c. Subjects must not have undergone autologous or allogeneic stem cell transplantation.

   d. Subjects must have initiated systemic therapy for multiple myeloma ≤1 year prior to physician-investigator confirmation of eligibility.

   e. Subjects must have achieved at least a minimal response (as defined by IMWG 2016 criteria1) to their overall systemic therapy for multiple myeloma and be clinically stable on their current regimen in the judgement of the investigator.
3. Subjects must not have achieved a stringent complete response according to IMWG 2016 criteria1 at time of physician-investigator confirmation of eligibility unless clonal plasma cells are detectable in bone marrow by flow cytometry (I.e., subjects in stringent complete response are eligible if minimal residual disease can be documented by bone marrow flow cytometry) or if residual disease is detectable by imaging such as PET/CT, CT, or MRI.
4. Subjects must have signed written, informed consent.
5. Subjects must be ≥ 18 years of age.
6. Subjects must have adequate vital organ function:

   1. Serum creatinine ≤ 2.5 or creatinine clearance ≥30 ml/min (measured or estimated according to CKD-EPI) and not dialysis-dependent.
   2. Absolute neutrophil count ≥1000/µl and platelet count ≥50,000/µl (≥30,000/µl if bone marrow plasma cells are ≥50% of cellularity).
   3. SGOT ≤ 3x the upper limit of normal and total bilirubin ≤ 2.0 mg/dl (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome).
   4. Left ventricular ejection fraction (LVEF) ≥ 45%. LVEF assessment must have been performed within 8 weeks of physician-investigator confirmation of eligibility.
7. Toxicities from prior/ongoing therapies, with the exception of peripheral neuropathy attributable to multiple myeloma therapy, must have recovered to grade ≤ 2 according to the CTCAE 5.0 criteria or to the subject's prior baseline.
8. Subjects must have an ECOG performance status of 0-2.
9. Subjects must be willing to forego first-line ASCT (Phase B and C patients only).
10. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in the protocol.

Exclusion Criteria:

1. Pregnant or lactating women
2. RETIRED WITH PROTOCOL V6
3. Active hepatitis B, hepatitis C, or HIV infection, or other active, uncontrolled infection.
4. Any uncontrolled medical or psychiatric disorder that would preclude participation as outlined.
5. NYHA Class III or IV heart failure, unstable angina, or a history of recent (within 6 months) myocardial infarction or sustained (>30 seconds) ventricular tachyarrhythmias.
6. Have active auto-immune disease, including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis, or have a history of severe (as judged by the physician-investigator) autoimmune disease requiring prolonged immunosuppressive therapy.
7. Have prior or active central nervous system (CNS) involvement (e.g. leptomeningeal disease, parenchymal masses) with myeloma. Screening for this (e.g. with lumbar puncture) is not required unless suspicious symptoms or radiographic findings are present. Subjects with calvarial disease that extends intracranially and involves the dura will be excluded, even if CSF is negative for myeloma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2036-03 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Adverse event reporting | 90 Days
  The occurrence of adverse events that are possibly, probably or definitely related to CAR T cells.

SECONDARY OUTCOMES:
Adverse event reporting | 15 years
  Occurrence of adverse events that are possibly, probably, or definitely related to study interventions during the primary or long-term follow-up phase.
Clinical outcomes after each CAR T cell regimen | 2 years
  Attainment of PET-negative response (absence of detectable FDG-avid disease by PET/CT).
Duration of Response | 15 years
  IMWG 2016 criteria will be used to define disease progression.
Progression-free Survival (PFS) | 15 years
  defined as time from initial CAR T cell until death or progression of multiple myeloma. IMWG 2016 criteria will be used to define disease progression.
Overall Survival (OS) | 15 years
Evaluate effects of huCART19 on correlative parameters of CART BCMA resistance and clonogenic multiple myeloma cells, such as the following: | 2 years
  Persistence of clonal BCMAdim/neg or CD19+ plasma cells as measured by flow cytometry and immunohistochemistry
  1. Depletion of multiple myeloma clonogenicity as measured using in vitro colony formation assays on bone marrow samples
  2. Induction of anti-Sox2 and other anti-myeloma immune responses
  3. Depletion of clonal CD19+ B cells
Composition of investigative products | 2 years
  Evaluate cellular composition of apheresis product and CARTBCMA/ huCART19 cells.
Maintenance therapy effects on persistence | 28 days post infusion - 2 years
  Evaluate effects of post-infusion maintenance therapy on CAR T cell persistence using quantitative molecular methods.
In vivo CAR T cell expansion as measured by flow cytometry | 28 days post infusion - 2 years
In vivo CAR T cell expansion as measured by qPCR | 28 days post infusion - 2 years
Duration of in vivo persistence of CAR T cells. | 28 days post infusion - 2 years
  As measured by flow cytometry and/or qPCR for vector sequences. For each parameter, CART-BCMA and huCART19 pharmacokinetics will be analyzed separately for patients receiving both products
Effects of maintenance therapy on CAR T cell pharmacokinetic parameters. | 28 days post infusion - 2 years
  As measured by flow cytometry and/or qPCR for vector sequences. For each parameter, CART-BCMA and huCART19 pharmacokinetics will be analyzed separately for patients receiving both products
Bioactivity by multiplex cytokine analysis | 28 days post infusion - 2 years
  As measured by flow cytometry and/or qPCR for vector sequences. For each parameter, CART-BCMA and huCART19 pharmacokinetics will be analyzed separately for patients receiving both products
Cellular composition of CAR T cell products | 28 days post infusion - 2 years
  cell-surface immunophenotype
Immune cell phenotyping | 2 years
  Characterize the cellular phenotype of multiple myeloma cells that persist after CAR T cell treatment using qualitative molecular methods.
Impact of T Cells on systemic soluble immune factors in patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Garfall, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Univ. of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Zhang Z, Markmann C, Yu M, Agarwal D, Rostami S, Wang W, Liu C, Zhao H, Ochoa T, Parvathaneni K, Xu X, Li E, Gonzalez V, Khadka R, Hoffmann J, Knox JJ, Scholler J, Marcellus B, Allman D, Fraietta JA, Samelson-Jones B, Milone MC, Monos D, Garfall AL, Naji A, Bhoj VG. Immunotherapy targeting B cells and long-lived plasma cells effectively eliminates pre-existing donor-specific allo-antibodies. Cell Rep Med. 2023 Dec 19;4(12):101336. doi: 10.1016/j.xcrm.2023.101336. PMID 38118406